CLINICAL TRIAL: NCT04840290
Title: A Neoadjuvant Study of Sintilimab Plus Platinum Doublet Chemotherapy in IIIA(N2) Stage Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Neoadjuvant Study of Sintilimab Plus Platinum Doublet Chemotherapy in IIIA(N2) Stage NSCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Yang Song, MD, Professor, Tang-Du Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCL201902
Record Dates: First submitted 2021-03-30; First posted 2021-04-09 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Neoadjuvant Study; Sintilimab; Stage IIIA (N+); NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Injections; Carboplatin

STUDY DESIGN:
Intervention Model Description: Sintilimab Plus Paclitaxel (Albumin Bound) and Platinum Doublet Chemotherapy in Stage of IIIA NSCLC, as the Neoadjuvant treatment.
Masking Description: this is a single-arm study, masking is not require.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab Plus Platinum Doublet Chemotherapy (Experimental): Specified dose on specified days Sintilimab
  Interventions: Drug: Biological: Sintilimab Drug: Cisplatin Drug: Paclitaxel for Injection (Albumin Bound) Drug: Carboplatin

INTERVENTIONS:
Drug: Biological: Sintilimab Drug: Cisplatin Drug: Paclitaxel for Injection (Albumin Bound) Drug: Carboplatin — Biological: Sintilimab Drug: Cisplatin Drug: Paclitaxel for Injection (Albumin Bound) Drug: Carboplatin

SUMMARY:
The purpose of this study is to determine the feasibility and evaluate the safety of delivering chemotherapy, the usual approach to non-small cell lung cancer, in combination with Sintilimab (PD-1 antibody), followed by adjuvant therapy after surgical resection. Consolidation therapy is treatment given following the initial treatment.

Sintilimab is an investigational drug, which has been approved by the NMPA(National Medical Products Administration,China. https://www.nmpa.gov.cn/) for use in late stage of non-small cell lung cancer (NSCLC). Sintilimab is a monoclonal antibody that binds to the surface of some cells of the immune system and activates them against cancer cells. It is not chemotherapy.

DETAILED DESCRIPTION:
The primary hypothesis is that the addition of Sintilimab to neoadjuvant concurrent chemotherapy, followed by consolidation Sintilimab, will be safe and feasible to deliver to patients with resectable stage 3A Non-small cell lung cancer (NSCLC).

This study also plans to observe the efficacy of this combination in the overall and biomarker-positive population.

Study Design This is an open-label, single arm phase III trial of neoadjuvant chemotherapy + Sintilimab with concurrent radiation followed by surgical resection and consolidation Sintilimab in resectable stage 3A (N2+) NSCLC.

Eligible patients will have biopsy-confirmed T1-3N2M0 (stage IIIA) non-small cell lung cancer (adenocarcinoma, squamous cell carcinoma, or large cell/NSCLC not otherwise specified), performance status 0-1, adequate lung function and deemed medically resectable by a thoracic surgeon, adequate organ function for chemotherapy, and no contraindications to Sintilimab (i.e. autoimmune disorders or underlying pulmonary fibrosis).

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed stage IIIA Non-Small Cell Lung Cancer without ALK，EGFR or ROS1 sensitive mutation Be willing and able to provide written informed consent/assent for the trial Have measurable or unmeasurable disease based on RECIST 1.1. Be willing to provide archival tissue from a tumor lesion or obtain a new biopsy if tissue unavailable.

Have a performance status of 0 or 1 on the Eastern Cooperative Oncology group (ECOG) Performance Scale.

Demonstrate adequate organ function Absolute neutrophil count (ANC) ≥1,500/mcL Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or erythropoiesis dependency Serum creatinine or Measured or calculated creatinine clearance ≤1.5 X upper limit of normal (ULN) or ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Serum total bilirubin ≤ 1.5 X ULN, or Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN Aspartate transaminase (AST) (SGOT) and Alanine transaminase (ALT) (SGPT) ≤ 2.5 X ULN or ≤ 5 X ULN for subjects with liver metastases Albumin ≥2.5 mg/dL International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

Presence of locally advanced, inoperable or metastatic disease Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment Has a known history of active Bacillus Tuberculosis (TB) Hypersensitivity to Sintilimab or any of its excipients. Has had any prior chemotherapy, targeted small molecule therapy, or radiation therapy for the currently diagnosed cancer.

Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.

Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

Has known history of, or any evidence of active, non-infectious pneumonitis. Has an active infection requiring systemic therapy. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.

Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies). Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C. Has received a live vaccine within 30 days of planned start of study therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 12 weeks after first day of neoadjuvant therapy
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
R0 Resection Rate | 12 weeks after first day of neoadjuvant therapy (day of surgery)
  Proportion of patients with complete tumor removal (R0 resection)

SECONDARY OUTCOMES:
Pathologic Complete Response Rate（pCR） | 12 weeks after first day of neoadjuvant therapy (day of surgery)
  Pathological complete response is defined as absence of foci of tumor cells at the local site (pCR)
Major Pathologic Responses Rate（MPR） | 12 weeks after first day of neoadjuvant therapy (day of surgery)
  The major pathologic response to preoperative therapy, defined histopathologically by the presence of less than 5% viable cancer cells in the surgical specimen, is an important prognostic factor for patients with NSCLC. In this study, we will calculate the proportion of patients with Major Pathologic Responses.
Complete Remission Rate | 12 weeks after first day of neoadjuvant therapy (day of surgery)
  the proportion of patients with disappearance of all signs of cancer in response to treatment. Also called complete response rate.
Progression Free Survival（PFS） | Up to approximately 69 months after the first disease progression
  Time from beginning of treatment to progression, death, or five years, whichever came first. Progression is defined as Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm
Overall Survival（OS） | Up to approximately 193 months
  The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive. In a clinical trial, measuring the OS is one way to see how well a new treatment works.

CONTACTS AND LOCATIONS:
Overall Officials: YANG SONG, MD, Principal Investigator — Tang-Du Hospital
Locations (1):
- TangDu hospital, the Airforce Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No